CLINICAL TRIAL: NCT06039462
Title: Improve Patient Safety and Wellbeing in Leeds Children Hospital for Patients Undergoing Procedures Through Use of Virtual Reality Distraction Therapy (VRDT), and Improve Their Overall Experience.
Brief Title: Virtual Reality Distraction Therapy in Paediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA21/140676
Record Dates: First submitted 2023-08-21; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children undergoing surgery (Other)
  Interventions: Behavioral: Application of a virtual reality headset

INTERVENTIONS:
Behavioral: Application of a virtual reality headset — Use of a headset to experience a different reality

SUMMARY:
For many children in hospital, having blood tests or cannulation is a significantly distressing event physically, psychologically and emotionally. Use of distraction during invasive procedures is already common practice in paediatrics to improve the experience both for the child and parents. Use of Virtual Reality (VR) and VR Distraction Therapy (VRDT) is a relatively new concept, but has already shown promising results in studies.

"VR offers an interactive distraction technique, a contrast to the passive distraction of reading a book or playing games on a tablet … and [VR] is thought to alter pain perception and the child's interpretation of pain signals." (Cochrane Library - Virtual reality simulation for reducing pain in children).

The project aims to collect data about venepuncture, cannulation, long lines - qualitative and quantitative data - from children and parents. This studyl compares current standard practice with VR distraction therapy.

DETAILED DESCRIPTION:
Not all studies raise significant issues. Some studies may have straightforward ethical or other issues that can be identified and managed routinely. Others may present significant issues requiring further consideration by a REC, HRA, or other review body (as appropriate to the issue). Studies that present a minimal risk to participants may raise complex organisational or legal issues. You should try to consider all the types of issues that the different reviewers may need to consider.

VR companies do not recommend use of their headsets in children under 13 years of age. I do not anticipate including 8-12 year olds in the study causing any issues based on experience and advice from relevant experts (see below). In summary, the age cut off is borne of lack of evidence for long-term effects of VR on visual or brain development, rather than specific concerns or evidence existing to inform the age cut off.

Children's Hospital Colorado (US) use VR in children of 6 years and above. Speaking with their Associate Professor of Paediatrics, the age limitation is not derived from medical standards or concerns. They discussed with their Neurology department who agreed there is no age-specific concern that warrants the 12 year cut-off, and they also rely upon the professional expertise of Child Life Specialists who routinely screen toys and devices for age-appropriate application. They have used VR in healthcare for children several hundred times and have no concerns about the age cut off the VR companies suggest.

Stanford University School of Medicine (US) run the highest volume clinical VR therapy program in the US, with thousands of children each year receiving VR. Their department similarly does not exclude under 13 year olds from their program.

Clinicians experienced with VR in the UK have spoken to VR companies involved in their studies, and the information gives was that there no long-term data on VR and its effects on brain and visual development. These clinicians also use VR on children aged 5-6 years and above.

I have met with the VR company Dubit Limited, which shows in its global trends data that children much younger than 13 are already using VR. The publication "Children and Virtual Reality: Emerging Possibilities and Challenges" contains data from studies looking at the 8-12 year old age group; there is not any current evidence of adverse events in this age group, though transient change to visual function has been seen only in a minority of VR users in this age group.

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric patient, aged 8-12 years or 13-18 years.
2. Under care of paediatric department - as inpatient
3. Requiring invasive procedure - including (but not limited to) blood sampling (venepuncture), siting intravenous access (cannulation, long line, Port-a-cath access), lumbar puncture, other device insertion or removal (e.g. catheter, drain, cardiac pacing wires, intra-thecal baclofen pump refills), minor surgical bedside procedures.
4. Consents to study - either child with mental capacity, or parent/legal guardian on behalf of their child.

Exclusion Criteria:

* Participants will not be recruited if they or their parent/guardian believe the child will not engage or cannot engage with procedural distraction.

Participants will not be recruited to the VR group if he/she meets any of the following exclusion criteria:

* Patients not under care of paediatrics (over 18 years of age)
* If the child has previously been recruited to the study - each child may only be in the study once
* Contraindications to use of VR or the VR headset

  * Inability to wear headset - facial or skull injury/fracture
  * Marked reduced visual acuity or blindness
  * Interference with care - e.g. requirement of other medical equipment that cannot be worn/administered simultaneously with VR e.g. non-invasive ventilation.
  * Pre-procedure dizziness, nausea, vertigo
  * History of photosensitive epilepsy
  * Potential for poor cooperation with procedure (hence risk of moving) - this is more likely in the age range 8-12 years old. Prior discussion to be held with parents through PIL and consent form to judge if the child is likely to be cooperative.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Reduction in fear and anxiety associated with treatment. | 24 hours
  Questionnaire (x1) completed at the time of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hopsital NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No